CLINICAL TRIAL: NCT07271667
Title: A Phase 2 Study of Emavusertib in Combination With an Approved Bruton Tyrosine Kinase Inhibitor in Patients With Chronic Lymphocytic Leukemia and Other B-cell Malignancies
Brief Title: A Study of Emavusertib + An Approved Bruton Tyrosine Kinase Inhibitor (BTKi) in Participants With Chronic Lymphocytic Leukemia (CLL) and Other B-cell Malignancies
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA-4948-203; 2025-523600-68-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; B-cell Malignancies
Keywords: Emavusertib; BTKi; B-cell Malignancies; Chronic Lymphocytic Leukemia; CLL; Zanubrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Emavusertib and Zanubrutinib (Experimental): Participants in Cohort 1 include CLL participants who have been on zanubrutinib for at least 12 months and are currently in a partial response (PR) or partial response with lymphocytosis (PR-L) and measurable residual disease positive (MRD+). In Part A, participants will receive one of two doses of emavusertib twice daily (BID) and an approved dose of zanubrutinib per label. In Part B, additional participants will be enrolled in an expansion if pre-defined criteria for Part A are met. Participants will receive one of two doses of emavusertib BID and an approved dose of zanubrutinib per label.
  Interventions: Drug: Emavusertib; Drug: Zanubrutinib
- Cohort 2: Emavusertib and Zanubrutinib (Experimental): Participants in Cohort 2 include relapsed CLL participants who have directly progressed on zanubrutinib after a confirmed response (PR or better lasting 6 months or longer). In Part A, participants will receive one of two doses of emavusertib BID and an approved dose of zanubrutinib per label. In Part B, additional participants will be enrolled in an expansion if pre-defined criteria for Part A are met. Participants will receive one of two doses of emavusertib BID and an approved dose of zanubrutinib per label.
  Interventions: Drug: Emavusertib; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Emavusertib — Oral tablets
Drug: Zanubrutinib — Oral capsules
  Other Names: BRUKINSA®

SUMMARY:
The primary objective of the study for Cohort 1 and Cohort 2 is to assess the anticancer activity of emavusertib in combination with zanubrutinib in participants with CLL.

ELIGIBILITY:
Inclusion Criteria (All Parts):

1. Males and females ≥ 18 years of age.
2. Life expectancy of ≥ 3 months.
3. Eastern Cooperative Oncology Group Performance Status of 0, 1, or 2.
4. Histopathologically confirmed diagnosis of CLL (medical record is acceptable), as per the World Health Organization 2016 classification.
5. At least 1 criterion for measurable disease per International Workshop on Chronic Lymphocytic Leukemia (iwCLL).
6. For Cohort 1 only:

   1. Participant must be in a partial response (PR) or partial response with lymphocytosis (PR-L) and measurable residual disease positive (MRD+) per Hallek et al, (2018) criteria.
   2. Participant must have detectable measurable residual disease (MRD) as determined by the ClonoSEQ assay
   3. Must be actively taking zanubrutinib for at least 12 months.
   4. Acceptable organ function at Screening within 28 days prior to Cycle 1 Day 1 (C1D1)
7. For Cohort 2 only:

   1. Relapsed disease for which participants are ineligible for or have exhausted standard therapeutic options that would be considered standard of care
   2. Must be actively taking zanubrutinib.
   3. Participants must have had direct progression on zanubrutinib (within 3 months prior to study entry; administered as monotherapy or in combination) and no other anticancer therapy administered since.
   4. Acceptable organ function at Screening within 28 days prior to C1D1.
8. Creatine phosphokinase (CPK) < 2.5 × ULN.
9. Ability to tolerate a contrast-enhanced computed tomography (CT) scan.
10. Ability to swallow and retain oral medications.
11. Negative serum pregnancy test in women of childbearing potential (WOCP).
12. WOCP and men who partner with WOCP must agree to use highly effective contraceptive methods for the duration of the study and for 180 days after the last dose of study treatment.
13. Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria (All Parts):

1. Active second malignancy unless in remission with a life expectancy of > 2 years and with documented Sponsor approval.
2. Active malignancy other than CLL requiring systemic therapy (exceptions may be granted following a discussion with the Sponsor Medical Monitor).
3. Have high-risk CLL TP53 mutations and 17P deletion.
4. History of Grade ≥ 3 rhabdomyolysis without complete recovery.
5. Received prior chimeric antigen receptor-T cell therapy.
6. Received prior investigational drugs (including treatment in clinical research, unapproved combination products, and new dosage forms) within 28 days or 5 half-lives, whichever is shorter, prior to C1D1; allogeneic hematopoietic stem cell transplant (HSCT) within 60 days prior to C1D1; or had clinically significant graft-versus-host disease (GVHD) requiring ongoing uptitration of immunosuppressive medications prior to Screening.
7. Any prior systemic anticancer treatment such as chemotherapy, immunomodulatory drug therapy, etc., received within 21 days or 5 half-lives, whichever is shorter, prior to C1D1 (with the exception of zanubrutinib, which may be continued until the day before C1D1).
8. Receiving the following medications within 7 days or 5 half-lives, whichever is shorter, prior to C1D1:

   1. Medications that, in the opinion of the Investigator, have a high risk of causing prolonged QT interval, corrected (QTc) and/or Torsades de Pointes.
   2. Peg-filgrastim or equivalent.
   3. St John's Wort.
9. History of or ongoing drug-induced pneumonitis.
10. History of stroke or intracranial hemorrhage within 6 months prior to C1D1. Participants with post-biopsy hemorrhagic sequela defined as a small hyperdense lesion < 3 millimeters (mm) on T2 sequence will not be excluded.
11. Requirement for anticoagulation with warfarin or equivalent vitamin K antagonists, including dual antiplatelet agents, within 5 half-lives of the anticoagulant or 7 days, whichever is longer, prior to C1D1. Low molecular weight heparin is allowed. Participants who require the use of antiplatelet agents should be discussed with the Sponsor Medical Monitor (e.g., use of factor Xa inhibitors).
12. Vaccinated with a live-attenuated vaccine within 4 weeks prior to C1D1.
13. Prior history of hypersensitivity or anaphylaxis to emavusertib, zanubrutinib, or any of their excipients.
14. Prior history of Stevens-Johnson syndrome or toxic epidermal necrolysis.
15. Intolerance to contrast-enhanced CT scan due to allergic reactions to contrast agents.
16. Major surgery < 28 days prior to C1D1; minor surgery < 7 days prior to C1D1.
17. Viral infections:

    1. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome (AIDS)-related illness. If HIV is undetectable or maintained on treatment, enrollment may be allowed after discussion with the Sponsor Medical Monitor.
    2. Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive or hepatitis C virus (HCV) infection < 6 months prior to C1D1, unless viral load is undetectable, or HCV with cirrhosis.
    3. Active systemic infection, including HIV, cytomegalovirus infection, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, or has had, within 28 days prior to C1D1, an infection (other than nail trichophytosis) that requires hospitalization or an intravenous antibiotic.
18. Concomitant illness that would preclude safe participation in the study.
19. Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Undetectable Measurable Residual Disease (uMRD) Rate | Up to approximately 23 months
Cohort 2: Overall Response Rate (ORR) | Up to approximately 23 months

SECONDARY OUTCOMES:
Cohort 1: Duration of uMRD | Up to approximately 23 months
Cohort 1: Time to Measurable Residual Disease (MRD) Conversion | Up to approximately 23 months
Cohort 1: Complete Response (CR) Rate | Up to approximately 23 months
Cohort 1: Duration of CR | Up to approximately 23 months
Cohort 1: Time to CR | Up to approximately 23 months
Cohort 2: Duration of Response (DOR) | Up to approximately 23 months
Cohort 2: Time to Response | Up to approximately 23 months
Cohorts 1 and 2: Progression-free Survival (PFS) | Up to approximately 23 months
Cohorts 1 and 2: Overall Survival (OS) | Up to approximately 23 months
Cohorts 1 and 2: Number of Participants with Treatment-emergent Adverse Events (TEAEs) and Treatment-related Adverse Events | Up to approximately 23 months
Cohorts 1 and 2: Maximum Plasma Concentration (Cmax) of Emavusertib and Zanubrutinib | Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle = 28 days)
Cohorts 1 and 2: Time to Maximum Concentration (Tmax) of Emavusertib and Zanubrutinib | Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle = 28 days)
Cohorts 1 and 2: Area Under the Curve (AUC) from 0 to t Hours (AUC0-t) of Emavusertib and Zanubrutinib | Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle = 28 days)
Cohorts 1 and 2: Trough Plasma Concentration (Cmin) of Emavusertib and Zanubrutinib | Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle = 28 days)

IPD SHARING:
Plan to Share IPD: No